CLINICAL TRIAL: NCT04677855
Title: A Phase I Study of PCUR-101 in Combination With Androgen Directed Therapy in the Treatment of Patients With Metastatic Castration-Resistant Prostate Cancer
Brief Title: Study of PCUR-101 in Combination With ADT in Patients With mCRPC
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Business Decision due to insufficient enrollment
Sponsor: Pellficure Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PCUR101-003
Record Dates: First submitted 2020-12-14; First posted 2020-12-21 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Dutasteride; abiraterone; Prednisone

STUDY DESIGN:
Intervention Model Description: Part 1 dose escalation followed by a dose expansion
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- PCUR-101 Dose Escalation (Experimental): PCUR-101 dosed orally once per day in 28 day cycles. Patients will be enrolled into escalating dose levels during the dose escalation phase
  Interventions: Drug: PCUR-101
- PCUR-101 Dose Expansion Cohort 1 (Experimental): PCUR-101 dosed orally once per day in 28 day cycles
  Interventions: Drug: PCUR-101
- PCUR-101 Dose Expansion Cohort 2 (Experimental): PCUR-101 in combination with dutasteride dosed orally once per day in 28 day cycles
  Interventions: Drug: PCUR-101; Drug: Dutasteride 0.5 mg
- PCUR-101 Dose Expansion Cohort 3 (Experimental): PCUR-101 dosed orally once per day in combination with abiraterone (once per day) and prednisone (twice per day) in 28 day cycles
  Interventions: Drug: PCUR-101; Drug: Abiraterone and Prednisone

INTERVENTIONS:
Drug: PCUR-101 — 50 mg capsules
Drug: Dutasteride 0.5 mg — 0.5 mg capsules
  Arms: PCUR-101 Dose Expansion Cohort 2
Drug: Abiraterone and Prednisone — 500 mg tablets Abiraterone with 5 mg Prednisone Tablets
  Arms: PCUR-101 Dose Expansion Cohort 3

SUMMARY:
This is an open label, non-randomized, Phase I, dose escalation/dose expansion study in cohorts of patients with metastatic CRPC at Screening. Dose escalation uses a 3+3 design to determine the maximum tolerated dose (MTD). Once the MTD is defined, the dose expansion phase is used to define the recommended phase 2 dose.

DETAILED DESCRIPTION:
Dose Escalation Phase: Eligible patients will enter the study and start receiving daily doses of PCUR-101 during Cycle 1. Subsequent dose cohorts will receive the next higher dose of PCUR-101 according to a 3 + 3 design until the MTD is determined. Patients may remain on these treatment cycles if they do not progress or experience any dose limiting toxicities (DLTs).

Dose Expansion Phase: Once the MTD has been determined, approximately 18 patients in 3 cohorts will be enrolled for further evaluations of safety, PK, and preliminary clinical activity during successive 28-day cycles in the dose expansion phase: Expansion Cohort 1 will receive PCUR-101 at the MTD, Expansion Cohort 2 will receive PCUR-101 at one dose level lower than the MTD and dutasteride once daily, and Expansion Cohort 3 (6 patients) will receive PCUR-101 at one dose level lower than the MTD in patients about to start abiraterone (1000 mg QD) and prednisone (5 mg twice daily [BID]) as their standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of prostate cancer
* Demonstrates metastatic CRPC
* Castrate level of serum testosterone at screening
* Adequate hematologic, renal, and hepatic function
* ECOG status ≤1
* Life expectancy of at least 3 months
* No more than one prior course of cytotoxic chemotherapy

Exclusion Criteria:

* Pure small cell, neuroendocrine or other variant (non-adenocarcinoma) prostate cancer histology
* Visceral metastasis excluding lymph nodes
* Use of opiate analgesics for prostate cancer pain or non-cancer pain
* other investigational agents or concurrent anticancer therapy other than standard androgen deprivation therapy within 4 weeks
* History of bleeding disorder
* History of seizure disorder
* Concomitant use of warfarin
* Prior exposure to PCUR-101
* History of myocardial infarction, arterial thrombotic events, heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmia
* Received wide-field external beam radiation therapy within 4 weeks
* Moderate to severe neuropathy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2021-03-30 (Actual); Primary Completion 2023-10-23 (Actual); Study Completion 2023-11-20 (Actual)

PRIMARY OUTCOMES:
Occurrence of Dose Limiting Toxicity | over the first 28 days of dosing
  Incidence of Adverse Adverse Events

SECONDARY OUTCOMES:
Determination of pharmacokinetic parameters - Tmax | over the first 28 days of dosing
  time to peak concentrations of PCUR-101
Determination of pharmacokinetic parameters - Cmax | over the first 28 days of dosing
  peak concentrations of PCUR-101
Determination of pharmacokinetic parameters - T1/2 | over the first 28 days of dosing
  time from maximum concentration PCUR-101 to a reduction of plasma concentration by 50%
Preliminary Evidence of efficacy/anti tumor activity - PSA levels | through study completion, average of 12 months
  as assessed by PSA changes
Preliminary Evidence of efficacy/anti tumor activity - RECIST | through study completion, average of 12 months
  as assessed by RECIST 1.1 criteria

CONTACTS AND LOCATIONS:
Locations (4):
- United States (2):
  - University of Michigan, Ann Arbor, Michigan
  - Nebraska Cancer Specialist, Omaha, Nebraska
- Australia (2):
  - St. George Private Hospital, Kogarah, New South Wales
  - Southern Oncology Clinical Research, Bedford Park, South Australia

IPD SHARING:
Plan to Share IPD: No